CLINICAL TRIAL: NCT00195949
Title: Laparoscopic Versus Open Pyloromyotomy for Infants With Idiopathic Hypertrophic Pyloric Stenosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-01-004
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2005-09

CONDITIONS: Hypertrophic Pyloric Stenosis
Keywords: Pyloric Stenosis; Laparoscopy; Idiopathic Hypertrophic Pyloric Stenosis
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic; Pyloric Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Laparoscopic pyloromyotomy

SUMMARY:
Pyloric stenosis is a condition that develops in infants and that leads to an obstruction of the channel going out of the stomach. This study is being performed to determine if there is an advantage to the laparoscopic approach or the open approach for the surgical correction of the enlarged pylorus.

DETAILED DESCRIPTION:
Pyloromyotomy for pyloric stenosis has traditionally been performed via an open technique. With advancements in minimally invasive surgery in infants a laparoscopic approach has been developed. These two approaches have never been critically evaluated with regard to superiority of one technique over the other. This is a prospective randomized trial involving infants with pyloric stenosis. It will enroll 100 patients in each arm (statistical and power analysis was performed by Steve Simon, PhD). Parental consent will be obtained and the patients will be randomized to undergo open or laparoscopic pyloromyotomy. Patient age at diagnosis, electrolyte disturbances at diagnosis, ultrasound findings, operative approach, length of pyloromyotomy, operative times, time to tolerating full feeds, number of emesis episodes, length of hospitalization, operative charges, and hospital charges will be collected for comparison between the groups.

ELIGIBILITY:
Inclusion Criteria:

* All infants less than 12 weeks of age who have undergone surgical consultation and abdominal ultrasound confirming the diagnosis of pyloric stenosis and whose parents have given consent for inclusion in the study.

Exclusion Criteria:

* All patients greater than 12 weeks of age, or without parental consent, or without pyloric stenosis will be excluded from the study.

Max Age: 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200
Dates: Start 2003-04; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Operative Time

SECONDARY OUTCOMES:
Time to full feeds
Length of hospitalization
Pain medication requirements
Emesis episodes
Complications

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Ostlie, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States